CLINICAL TRIAL: NCT00005666
Title: Utility of Anatometabolic Imaging for Radiation Treatment Planning for Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1662; M01RR000042 (NIH)
Record Dates: First submitted 2000-05-19; First posted 2000-05-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Diagnostic imaging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Procedure: PET scan use in radiotherapy planning

SUMMARY:
This is a research study for patients with inoperable lung cancer called non-small cell lung cancer (NSCLC). Currently, the information from a radiological test, computed tomography (CT) scan of the chest, is used to design the best arrangement of radiation beams which will kill tumor cells and still spare the normal parts of lungs and other normal organs in the chest. The purpose of this study is to explore whether adding information from another radiological test, called positron emission tomography (PET), will improve the accuracy of the radiation beam arrangement designed to treat lung cancer. A PET scan is a way to picture the biochemistry of tissues and organs: of how tissues in the body take up glucose, a normal nutrient of the body. The researchers will attempt to create radiation treatment plans from PET images alone and compare differences between hypothetical plans and standard-of-care CT-based radiation treatment plans. Because there is honest uncertainty about the contribution of PET to radiation treatment planning, it is possible that there will be no difference between a CT-based treatment plan and one resulting from PET information. It is also possible that the addition of PET may result in a radiation beam arrangement that may better control lung cancer. The addition of PET may also result in treating less normal tissues, which may lower the risk of radiation side effects. This study will provide the preliminary data necessary to design a larger clinical trial that may define the role of PET in radiation treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced NSCLC (squamous, large cell undifferentiated or adenocarcinoma).
* Disease limited to the thorax, adjacent mediastinum and neurovascular structures, and supraclavicular or scalene lymph node area, as defined by the AJCC Staging System. This includes patients with Stage IIIA and IIIB disease.
* Performance status of 0-2 by Southwest Oncology Group criteria.
* Medically inoperable patients (Stage I or II)
* Locoregional recurrent tumor following surgery will be eligible provided they meet other eligibility criteria.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- UH B2 C490 Box 0010 E. Medical Center Drive, Ann Arbor, Michigan, United States